CLINICAL TRIAL: NCT04694625
Title: Effects of Structured Rehabilitation Program on Pain and Function in Patients With Total Knee Replacement
Brief Title: Structured Rehabilitation Program for Patients With Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/20/1041/M. Arsalan
Record Dates: First submitted 2021-01-03; First posted 2021-01-05 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Knee
Keywords: Knee pain; knee Replacement; Degenerative knee disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured rehabilitation program (Experimental): Structured rehabilitation program & conventional physical therapy
  Interventions: Other: Structured Rehabilitation Program; Other: Conventional Physical Therapy
- conventional physical therapy (Active Comparator): conventional physical therapy
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Structured Rehabilitation Program — Early Function Phase (Protective phase) week 1 Progressive Function Phase (Recovery Phase) 2nd and 3rd week Advance Function Phase (Activity Phase) 4th week
  Arms: Structured rehabilitation program
Other: Conventional Physical Therapy — • Rapid post-operative mobilization • Range of motion exercises started • Passive extension by placing pillow under foot • Flexion-by dangling the leg over the side of bed • Muscle strengthening exercises • Weight bearing is allowed on 1st post-operative

SUMMARY:
This study will be a randomized controlled trial. This study will be conducted in Horizon Hospital Lahore. A sample size of 26 patients will be taken. Patients will be divided into two groups by lottery method. Group A will be treated with Structured Rehabilitation program along with conventional physiotherapy while Group B will be treated with conventional physiotherapy only. Both groups will receive treatment for 4 weeks,3 sessions per week. The outcome measures Numeric pain rating scale(NPRS),6 minutes' walk test and Womac scale will be measured at baseline and at the end of 4th week. Data will be analyzed by SPSS 25.

DETAILED DESCRIPTION:
Total knee replacement (TKR) is the most common, gold standard surgical intervention in relieving pain, improving physical functions and quality of life in end-stage osteoarthritis.An estimated 25-47% of patients who are eligible for primary joint replacement in the United Kingdom have isolated unicompartmental osteoarthritis, and would be eligible to receive either implant.

Adequate post-operative pain control in TKR patients is very important as inadequate pain control can lead to delayed mobilization, prolonged hospital stay, deep vein thrombosis with embolic events, increased psychological stress thereby increasing morbidity and mortality of TKR patients.Physiotherapy, principally exercise prescription and gait re- education, is advocated for people after THR and TKR.Surgeons are particularly concerned regarding cementless implants, given they rely on press fit fixation in the surrounding bone for primary stability.Patients undergoing total knee arthroplasty often have unfulfilled expectations from the surgery that can lead to dissatisfaction.Patients have a poor understanding of outcomes related to total knee replacement (TKR) surgery, with most patients underestimating the potential benefits and overestimating the risk of complications.To prevent chronic pain after TKR, several perioperative interventions show benefits and merit further research. Enhanced Recovery After Surgery (ERAS) has been successfully adopted across a range of procedures with using rehabilitation program. This study will focus on effects of structured rehabilitation program of 4 weeks with different goals in each week for reducing pain and improving function in patients with knee osteoarthritis. Study will provide a structured rehabilitation program for the physiotherapist to achieve all goals in three phases (protective, Recovery & Activity phase).

AP Antony-Leo 2019 in this RCT study improvements occurred by following structured rehabilitation care,quality of life and joint specific outcomes through medial parapatellear approach.Andrew David Beswick. In TKR to prevent chronic pain, showing benefits by using several perioperative interventions.In this systematic review the patients with osteoarthritis achieve long term outcomes after TKR by using perioperative interventions. In evidence base review enhanced recovery after surgery had already been used successfully in various surgical specialities. This evidence-based review provides an insight into the best evidence linked to each component and their rationale for inclusion in the proposed enhanced recovery after surgery protocol. Arijit Goshi 2019. In this evidence base review enhanced recovery programmes require a multidisciplinary team of dedicated professionals, principally involving preoperative education, multimodal pain control and accelerated rehabilitation; this will be enhanced if combined with minimally invasive surgery. The current economic environment and restricted healthcare budget further necessitate brief hospitalisation while minimising costs.MS Ibrahim 2019.C.E.H Scott 2019. The patient satisfaction rate of 81.4 % at 12 month in this study is comparable to other studies.In this prospective study it is important to clear that whether dissatisfaction is a consequence of surgical technique, implant design, patient selection, or counselling and the management of expectation. This study provided knowledge about to help patient selection and counselling. Soren T.Sku 2019 in an RCT study in patients with knee osteoarthritis who were eligible for total knee replacement, treatment with total knee replacement followed by nonsurgical treatment resulted in greater pain relief and functional improvement after 12 month as compared to nonsurgical treatment.Literature shows that postoperative rehabilitation for total knee replacement is of prime importance and improves postoperative outcomes and it would be more beneficial to divide outcome goals in phases so as to achieve these goals according to week wise distribution

ELIGIBILITY:
Inclusion Criteria:

• Patient with unilateral or bilateral total knee replacement through medial parapatellar approach.

Exclusion Criteria:

* Patients awaiting revision TKR
* Post traumatic patients planned for TKR
* Those with non-degenerative joint diseases
* Patients got infected after operation

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4th week
  NPRS is a segmented version of Visual Analogue Scale (VAS). It consists of number from 0 to 10. Patient selects a number that best reflects his/her pain intensity where 0 is no pain and 10 is maximum pain. For construct validity, NPRS was highly correlated to Visual Analogue Scale (VAS) (0.86-0.95). The test-retest reliability of this scale is recorded to be 0.96. (Hawker et al. 2011)
6 Minute walk test | 4th week
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance (6 MWD) provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.
  The 6 MWT provides information regarding functional capacity, response to therapy and prognosis across a broad range of chronic cardiopulmonary conditions. Main strengths of the 6 MWT stem from its simplicity in concept and performance, low cost, ease of standardization, and acceptance by test subjects, including those who are deconditioned, elderly, or frail.
WOMAC SCALE | 4th week
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. The WOMAC measures five items for pain (score range 0- 20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).[2] Physical functioning questions cover everyday activities such as stair use, standing up from a sitting or lying position, standing, bending, walking, getting in and out of a car, shopping, putting on or taking off socks, lying in bed, getting in or out of a bath, sitting, and heavy and light household duties.

CONTACTS AND LOCATIONS:
Overall Officials: Saima Zahid, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Horizon Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antony-Leo AP, Arun-Maiya G, Mohan-Kumar M, Vijayaraghavan PV. Structured Total Knee Replacement Rehabilitation Programme and Quality of Life following Two Different Surgical Approaches - A Randomised Controlled Trial. Malays Orthop J. 2019 Jul;13(2):20-27. doi: 10.5704/MOJ.1907.004. PMID 31467647
- [Background] Willis-Owen CA, Brust K, Alsop H, Miraldo M, Cobb JP. Unicondylar knee arthroplasty in the UK National Health Service: an analysis of candidacy, outcome and cost efficacy. Knee. 2009 Dec;16(6):473-8. doi: 10.1016/j.knee.2009.04.006. Epub 2009 May 22. PMID 19464898
- [Background] Nussenzveig TC. Pain management after total joint replacement and its impact on patient outcomes. AORN J. 1999 Dec;70(6):1060-2. doi: 10.1016/s0001-2092(06)62213-8. No abstract available. PMID 10635429
- [Background] Skrejborg P, Petersen KK, Beck J, Ulrich M, Simonsen O, Nielsen PT, Arendt-Nielsen L, Laursen M. Investigating the Effect of Perioperative Chlorzoxazone on Acute Postoperative Pain After Total Hip and Knee Replacement Surgery. Clin J Pain. 2020 May;36(5):352-358. doi: 10.1097/AJP.0000000000000805. PMID 31977370
- [Background] Mohammad HR, Kennedy JA, Mellon SJ, Judge A, Dodd CA, Murray DW. The clinical outcomes of cementless unicompartmental knee replacement in patients with reduced bone mineral density. J Orthop Surg Res. 2020 Jan 31;15(1):35. doi: 10.1186/s13018-020-1566-2. PMID 32005197
- [Background] Levinger P, Bartlett JR, Bergman NR, McMahon S, Menz HB, Hill KD. The discrepancy between patient expectations and actual outcome reduces at the first 6 months following total knee replacement surgery. Knee Surg Sports Traumatol Arthrosc. 2019 Jul;27(7):2042-2050. doi: 10.1007/s00167-018-5210-1. Epub 2018 Oct 8. PMID 30298413
- [Background] Fraenkel L, Benjamin Nowell W, Stake CE, Venkatachalam S, Eyler R, Michel G, Peters E. Impact of Information Presentation Format on Preference for Total Knee Replacement Surgery. Arthritis Care Res (Hoboken). 2019 Mar;71(3):379-384. doi: 10.1002/acr.23605. PMID 29799668
- [Background] Beswick AD, Dennis J, Gooberman-Hill R, Blom AW, Wylde V. Are perioperative interventions effective in preventing chronic pain after primary total knee replacement? A systematic review. BMJ Open. 2019 Sep 6;9(9):e028093. doi: 10.1136/bmjopen-2018-028093. PMID 31494601
- [Background] Wainwright TW, Immins T, Antonis JHA, Taylor H, Middleton RG. Can the introduction of Enhanced Recovery After Surgery (ERAS) reduce the variation in length of stay after total ankle replacement surgery? Foot Ankle Surg. 2019 Jun;25(3):294-297. doi: 10.1016/j.fas.2017.12.005. Epub 2017 Dec 21. PMID 29409177
- [Background] Ghosh A, Chatterji U. An evidence-based review of enhanced recovery after surgery in total knee replacement surgery. J Perioper Pract. 2019 Sep;29(9):281-290. doi: 10.1177/1750458918791121. Epub 2018 Sep 13. No abstract available. PMID 30212288
- [Background] Ibrahim MS, Alazzawi S, Nizam I, Haddad FS. An evidence-based review of enhanced recovery interventions in knee replacement surgery. Ann R Coll Surg Engl. 2013 Sep;95(6):386-9. doi: 10.1308/003588413X13629960046435. PMID 24025284
- [Background] Scott CE, Howie CR, MacDonald D, Biant LC. Predicting dissatisfaction following total knee replacement: a prospective study of 1217 patients. J Bone Joint Surg Br. 2010 Sep;92(9):1253-8. doi: 10.1302/0301-620X.92B9.24394. PMID 20798443
- [Background] Skou ST, Roos EM, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen O, Rasmussen S. A Randomized, Controlled Trial of Total Knee Replacement. N Engl J Med. 2015 Oct 22;373(17):1597-606. doi: 10.1056/NEJMoa1505467. PMID 26488691
- [Background] Bade MJ, Struessel T, Dayton M, Foran J, Kim RH, Miner T, Wolfe P, Kohrt WM, Dennis D, Stevens-Lapsley JE. Early High-Intensity Versus Low-Intensity Rehabilitation After Total Knee Arthroplasty: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2017 Sep;69(9):1360-1368. doi: 10.1002/acr.23139. Epub 2017 Aug 13. PMID 27813347
- [Background] Barker KL, Beard D, Price A, Toye F, Underwood M, Drummond A, Collins G, Dutton S, Campbell H, Kenealy N, Room J, Lamb SE. COmmunity-based Rehabilitation after Knee Arthroplasty (CORKA): study protocol for a randomised controlled trial. Trials. 2016 Oct 13;17(1):501. doi: 10.1186/s13063-016-1629-1. PMID 27737685